CLINICAL TRIAL: NCT01236859
Title: Gabapentin for Prophylaxis Intrathecal Morphine-Induced Pruritus After Orthopedics Surgery
Brief Title: Gabapentin for Prophylaxis Intrathecal Morphine-Induced Pruritus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, maliwan oofuvong, Assistant Professor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GP180
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Pruritus
Keywords: Gabapentin; prophylaxis; incidence of pruritus; intrathecal morphine
MeSH Terms: conditions — Pruritus | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): The patients in the placebo group received equal numbers of identical looking placebo 2 h before operation
  Interventions: Drug: Gabapentin
- gabapentin (Active Comparator): Patients in the gabapentin group received two capsules of gabapentin 300 mg (Neurontin®, Pfizer) at 2 h before operation.
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Neurontin®, Pfizer
  Other Names: Neurontin®, Pfizer

SUMMARY:
Intrathecal morphine provides good postoperative analgesia for up to 18-24 hour after administration. Pruritus is the most common side effect of intrathecal morphine, which the incidence was reported as 20%-100%2 and 63% in Songklanagarind Hospital. Pathophysiology of opioid-induced pruritus remain unclear and more than one mechanism may be involved in the development of opioid-induced pruritus, such as, mediated central µ opioid receptors, Dopamine (D2) receptors, Serotonin (5-HT3) receptors, prostaglandin system, GABA receptors, and glycine receptors, so that why opioid-induced pruritus is difficult to manage. Many medications have been used to treat this side effect included antihistamines, 5-HT3 (serotonin) receptor antagonists, opioid antagonists, opioid agonist-antagonists, propofol, and nonsteroidal antiinflammatory drugs.

Gabapentin is an anticonvulsant, a structural analog of aminobutyric acid, and currently approved by the Food and Drug Administration for the treatment of partial seizures and postherpetic neuralgia. Many studies have shown gabapentin to be effective in the case of brachioradial pruritus, itch of neuropathic in origin, uremic pruritus, multiple sclerosis-induced pruritus,cholestatic pruritus, itch produced by burn, and pruritus of unknown origin. However, there is only one small study in Taiwan shown the effectiveness of gabapentin 1200 mg in prevention of intrathecal morphine-induced pruritus in orthopedic surgery, which could reduce incidence of pruritus from 77.5% to 47.5% (38.7% reduction). Because gabapentin has several side effects especially in high dose such as drowsiness, dry mouth, headache, unsteadiness, reduced co-ordination or slowed reaction, constipation, diarrhea, peripheral edema, dizziness, confusion, loss of concentration, weight gain, and nausea, vomiting, so in our study we decided to reduce the dose of gabapentin. Therefore, we would like to know if gabapentin in a smaller dose (600 mg) used in the wider range of age including the elderly can decrease the incidence of intrathecal morphine-induced pruritus in orthopedic surgery in Songklanagarind Hospital.

DETAILED DESCRIPTION:
The study was approved by the ethic committee of Songklanagarind Hospital in Songkhla, Thailand, and was designed as a randomized, double-blind, placebo-controlled trial. All patients gave their informed consent after receiving written information of the study. Orthopedic patients were invited to participated between September 2009 and August 2010. Patients were considered eligible if they were aged between 15-70 yr, ASA physical status I-III, and were scheduled for lower limb surgery under spinal anesthesia. Patients were excluded if they presented of any following reasons: contraindication for spinal anesthesia, known allergy history to gabapentin, complaint of pruritus before surgery, morbid obesity (BMI > 35), coexisting skin disorder, and any systemic disease associated with pruritus. Patients who had history of seizure attacks, mental illness, chronic headache, or neuropathic pain and were concomitantly using of anticonvulsants, antidepressants, antipsychotics, or antihistamine were also excluded. Patients were randomized into the treatment and the placebo groups according to a computer-generated randomization list and patients were allocated consecutively. The blinding was maintained by keeping the treatment code with one of the investigators, separating them from the investigator performing the assessments. Patients in the gabapentin group received two capsules of gabapentin 300 mg (Neurontin®, Pfizer) at 2 h before operation. The patients in the placebo group received equal numbers of identical looking placebo, according to the same schedule. In order to prepare the identical looking medications, for gabapentin group we coated gabapentin capsules by other capsules and for placebo group we filled the identical looking capsules with flour. All patients did not receive any other sedative agents beside the study drugs. After standard monitoring (electrocardiogram, noninvasive arterial blood pressure, and pulse oximetry) was set-up in the operating room, each patient was received Ringer's lactate or normal saline solution 5-10 mL/kg, spinal anesthesia was performed at the L2-3 or L3-4 interspace with a 27-gauge Quincke-type needle using 0.5% isobaric bupivacaine plus 0.2 mg of preservative-free morphine. Midazolam, morphine, fentanyl and propofol were administered intravenously (IV) for intraoperative sedation at the discretion of the anesthesiologist. We excluded the patient who failed spinal block, inadequate block, and the patient who had prolong operative time which had to continue with general anesthesia because we could not evaluate pruritus. The sedation level was evaluated by the Ramsay Sedation Scale during the operation. The patients were followed for 24 h after intrathecal administration of morphine. Postoperative wound pain was assessed with a verbal numeric rating scale (VNRS). Rescue treatments for postoperative pain were provided with any medications ordered by anesthesiologists or orthopedists. Pruritus was evaluated at 1, 2, 3, 4, 6, 9, 12, and 24 h after intrathecal administration of morphine by a blinded investigator. The patients were questioned about the presence and degree of pruritus. The degree of pruritus was classified as 0 = absent, 1 = mild (restricted to one area such as face or arms, not troubling the patient, often reported only after prompting), 2 = moderate (affecting a larger area such as face and arms or face and anterior surface of thorax, not disturbing the patient, therefore not requiring treatment), or 3 = severe (extensive or generalized, often disturbing the patient to the point of necessitating treatment). Severe pruritus was treated with 10 mg IV chlopheniramine. Patients were also evaluated the severity of postoperative nausea and vomiting (PONV) which graded on a four point scale as 0 = no nausea or vomiting, 1 = mild nausea only, 2 = nausea or vomiting responding to initial treatment, and 3 = nausea or vomiting requiring repeat treatment, the presence of urinary retention and the other side effects of drug treatment. Patients who reported vomiting received 4 mg IV ondansetron or 10 mg IV metoclopramide. The primary outcome measure of the study was the incidence of pruritus during the 24 h follow-up period. The difference of onset time and severity of pruritus in the gabapentin and placebo groups served as the secondary outcome measure. Additional secondary outcome measures were side effects of the gabapentin group. There was an intention-to-treat in our study. Statistical analysis was performed using the R 2.11.1 software. We considered a 35% reduction in the incidence of pruritus to be clinically important according to the previous study's result showed that gabapentin 1200 mg could reduce incidence of intrathecal morphine-induce pruritus by 38%12. In our study we reduced the dose of gabapentin to 600 mg as describe previously so we think the efficacy of the drug may decrease so we assumed that gabapentin 600 mg could reduced incidence of intrathecal morphine-induced pruritus by 35%. Power analysis was performed to determine the sample size with a probability for a type II error of 0.2 and type I error of 0.05. To detect a 35% reduction in the incidence of pruritus, using the incidence of pruritus in Songklanagarind Hospital which was 63%, a sample size of 80 patients in each group was estimated to be required. To accommodate for 10% patient dropouts and failure of spinal anesthesia, 88 patients were enrolled in each group. Incidence of pruritus was measured by using Chi-Square test. The onset time and severity of pruritus was analyzed by means of Kaplan-Meier probability curves. Continuous data were analyzed using un-paired student T-test for normal distribution data such as BMI and by Mann-Whitney U test for non normal distribution data such as age, operative time, postoperative verbal numeric rating pain score. Comparison of the categorical data was performed using chi-square test such as incidence of PONV, hypotension, and shivering and by Fisher's exact test if expected value < 5 such as type of operation, incidence of bradycardia, and ASA classification. Results are expressed as mean+SD for normal distribution data and median (range) for non normal distribution. For all determinations, P values of < 0.05 were considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* aged between 15-70 yr, ASA physical status I-III, and were scheduled for lower limb surgery under spinal anesthesia.

Exclusion Criteria:

* contraindication for spinal anesthesia, known allergy history to gabapentin, complaint of pruritus before surgery, morbid obesity (BMI > 35), coexisting skin disorder, and any systemic disease associated with pruritus. Patients who had history of seizure attacks, mental illness, chronic headache, or neuropathic pain and were concomitantly using of anticonvulsants, antidepressants, antipsychotics, or antihistamine

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
incidence of pruritus postoperatively | 0-24 h
  the incidence of pruritus during the 24 h follow-up period

SECONDARY OUTCOMES:
onset time and severity of pruritus | 0-24 h
  The difference of onset time and severity of pruritus in the gabapentin and placebo groups

CONTACTS AND LOCATIONS:
Overall Officials: Wirinda Chiravanich, MD, Principal Investigator — Prince of Songkhla University
Locations (1):
- Songklanagarind Hospital, Hat Yai, Changwat Songkhla, Thailand